CLINICAL TRIAL: NCT01508338
Title: The Effects of HMB, ATP, and HMB Plus ATP on Muscle Mass, Strength, and Power in Resistance Trained Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: University of Tampa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MTI2012-CS01
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Healthy Experienced Weight Training Males
Keywords: HMB beta-hydroxy-beta-methylbutyrate; ATP (adenosine-triphosphate); trained athletes
MeSH Terms: interventions — Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- HMB (Experimental)
  Interventions: Dietary Supplement: HMB
- ATP and HMB (Experimental)
  Interventions: Dietary Supplement: Peak ATP and HMB
- ATP (Experimental)
  Interventions: Dietary Supplement: ATP

INTERVENTIONS:
Dietary Supplement: Placebo — An oral placebo capsule will be taken each morning and three dosages of a placebo gel containing polydextrose will be taken 3 times daily for 12 weeks.
  Arms: Placebo
Dietary Supplement: HMB — A placebo capsule will be taken each morning and three dosages of HMB gel, each providing 1 g of HMB, will be taken daily for a total of 3 g HMB per day for 12 weeks.
  Arms: HMB
Dietary Supplement: Peak ATP and HMB — One capsule containing 400 mg of Peak ATP will be taken in the morning and three dosages of HMB gel, each providing 1 g of HMB, will be taken daily for a total of 3 g HMB per day for 12 weeks.
  Arms: ATP and HMB
Dietary Supplement: ATP — One capsule containing 400 mg of Peak ATP will be taken daily in the morning and three dosages of a placebo gel containing polydextrose will be taken 3 times daily for 12 weeks.
  Arms: ATP

SUMMARY:
The purpose of this study is to

* determine the effects of 12 weeks of HMB free acid gel, ATP, and HMB free acid gel plus ATP supplementation in trained individuals during a periodized training program on skeletal muscle hypertrophy, body composition, strength, force, velocity, and peak power during loaded and unloaded vertical jumps.

Additionally, the study will determine if either supplementation protocol prevents the typical decay seen in performance following an overreaching cycle performed in the 9th and 10th weeks of the study.

Finally, the study will elucidate the mechanisms of action of supplementation on protein breakdown by analyzing serum indices of muscle damage (CK, LDH) and anabolic status (Testosterone:Cortisol ratio) as well as a urinary indicator of protein breakdown (3-methylhistidine).

We hypothesize that under these conditions that the supplementation protocols will augment skeletal muscle hypertrophy, strength, and power and that HMB will blunt increases in serum indices of muscle damage, and urinary indices of protein breakdown.

DETAILED DESCRIPTION:
In a randomized and double blind study the subjects will consume either placebo supplements, HMB supplement, ATP supplement, or HMB plus ATP supplements for 12 weeks. While consuming the supplements the subjects will undergo an extensive resistance training program designed to train all major muscle groups. An additional overreaching training cycle during weeks 9 and 10 which will involve a high-volume, hypertrophy style training program.

Subject testing will consist of the following:

* Strength and power at weeks 0, 1, 4, 8, 9, 10, and 12
* Range of motion and muscle soreness at weeks 0, 1, 8, 9, and 10
* Body composition and muscle assessments at weeks 0, 1, 4, 8, 9, 10, and 12
* Body fat assessments at weeks 0, 4, 8, and 12
* Blood biochemical measurements at weeks 0, 1, 4, 8, 9, 10, and 12
* Urinary analysis for protein breakdown (3-methylhistidine) at 0, 1, 8, 9, and 10 weeks

ELIGIBILITY:
Subjects must meet all of the inclusion criteria to participate in the study.

* Have 3 years minimum of free weight training experience
* Can squat a minimum of 1.5 times their bodyweight
* Can bench press a minimum equal to their bodyweight
* Can deadlift a minimum of 1.5 times their bodyweight
* Are free of musculoskeletal injuries
* Have not taken creatine or HMB supplements for 6 weeks
* Are not taking amino acid supplements
* Are not using anabolic or catabolic hormones
* Are not taking medications that may interfere with study measurements
* Are not users of tobacco products

All candidates meeting any one of the exclusion criteria will not be enrolled into the study.

* Do not have 3 years minimum of free weight training experience
* Can not squat a minimum of 1.5 times their bodyweight
* Can not bench press a minimum equal to their bodyweight
* Can not deadlift a minimum of 1.5 times their bodyweight
* Are not free of musculoskeletal injuries
* Have not taken creatine or HMB supplements in the past 6 weeks
* Are currently taking amino acid supplements
* Are using anabolic or catabolic hormones
* Are taking medications that may interfere with study measurements
* Use of tobacco products

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Increased muscle strength, force, and power after intense weight training | 12 weeks

SECONDARY OUTCOMES:
Increased muscle hypertrophy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Study Director — Metabolic Technologies Inc.
Locations (1):
- University of Tampa, Tampa, Florida, United States

REFERENCES:
- [Derived] Wilson JM, Joy JM, Lowery RP, Roberts MD, Lockwood CM, Manninen AH, Fuller JC, De Souza EO, Baier SM, Wilson SM, Rathmacher JA. Effects of oral adenosine-5'-triphosphate supplementation on athletic performance, skeletal muscle hypertrophy and recovery in resistance-trained men. Nutr Metab (Lond). 2013 Sep 22;10(1):57. doi: 10.1186/1743-7075-10-57. PMID 24330670